CLINICAL TRIAL: NCT04347265
Title: Ultrasound-guided Neuromodulation Percutaneous in Lower Back Pain: a Pilot Study
Brief Title: Ultrasound-guided Neuromodulation Percutaneous in Lower Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Blanca de la Cruz Torres, Director, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NMP in lower back pain
Record Dates: First submitted 2020-04-12; First posted 2020-04-15 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Lower Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NMP in level 1 (Experimental): Participants in this group received NMP of the sciatic nerve in the gluteus region
  Interventions: Other: NMP
- NMP in level 2 (Experimental): Participants in this group received NMP of the sciatic nerve in the middle of the thigh
  Interventions: Other: NMP
- NMP in level 3 (Experimental): Participants in this group received NMP of the sciatic nerve before popliteus region
  Interventions: Other: NMP

INTERVENTIONS:
Other: NMP — Participants received the percutaneous electrical stimulation intervention. Specifically, this consisted of the application of a square wave biphasic electrical current, with 3 Hz frequency and a 250µs pulse width, at the maximal tolerable intensity, to cause an tolerable muscle contraction. The application was 10 stimulations of 10 seconds, with 10 seconds at rest between stimulations. A trained physiotherapist performed the PNM intervention.

SUMMARY:
In our daily clinical practice, one of the most frequent reasons for consultation physiotherapists is low back pain (LBP). Regardless of the origin of the problem, the approach from physiotherapy contemplates the reduction of pain through different procedures, including neuromodulation.

In the field of Physiotherapy, ultrasound-guided Percutaneous Neuromodulation (PNM) is defined as the application through a needle with ultrasound guidance of an electrical current at low or medium frequency, seeking a sensitive and / or motor response of a peripheral nerve in some point of its trajectory, or of a muscle in a motor point, with a therapeutic objective. The objective of this study is to analyze that the effect of PNM on the sciatic nerve produces statistically significant changes in pain, joint range and functionality in patients with chronic LBP. Thirty subjects will be recruited, which will be divided into 3 groups: group 1 to which PNM will be applied to the sciatic nerve in the gluteus region; group 2 to which PNM will be applied to the sciatic nerve in the middle of the thigh; and group 3 to which PNM will be applied to the sciatic nerve before popliteus region. The PNM intervention with NMP will consist in the single application of an asymmetric rectangular biphasic current (250 microseconds, 3 Hz) during 90 seconds

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Lower Back Pain
* Having no other therapy

Exclusion Criteria:

* Other pathology (discal hernia, injured limbs, neurological pathology)
* Belenophobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2020-05-09 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Level of pain | From baseline measurement up to 1 week
  Measured by Visual Analogue Scale (0, no pain; 100, max pain)
Range of motion | From baseline measurement up to 1 week
  Measured by goniometer. Hip flexion, external and internal rotation range of motion
Y Balance Test | From baseline measurement up to 1 week
  Stability body
Owestry questionnaire | From baseline measurement up to 1 week
  Lower back pain questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Blanca De la Cruz Torres, PhD, Study Director — University of Seville
Locations (1):
- Blanca de la Cruz Torres, Seville, Spain

IPD SHARING:
Plan to Share IPD: No